CLINICAL TRIAL: NCT04071548
Title: The Effect of Exercise on Muscle Dysfunction in Cystinosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Richard Reimer, Effect of exercise on muscle dysfunction in cystinosis, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46941
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Cystinosis
MeSH Terms: conditions — Cystinosis | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Single site interventional exercise study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIIT Exercise (Experimental): All individuals recruited in exercise portion will be on an active exercise intervention
  Interventions: Other: HIIT Exercise

INTERVENTIONS:
Other: HIIT Exercise — HIIT exercise bike protocol
  * 3 minute warm up
  * Intervals of 10x 60 sec of 80-95% of heart rate reserve Heart rate reserve = Max Heart rate - Resting Heart rate § Max heart rate = 220-age
  * 10x60 second Recovery period
  * 5 minute cool-down
  Other Names: High Intensity Interval Training

SUMMARY:
Classification of activity tolerance is of importance in chronic progressive myopathies, not only to better understand functional implications of the disease state itself, but also for purposes of exercise prescription for health maintenance. Maximal exercise testing has been considered as the gold standard of assessing maximal aerobic capacity, however testing in individuals with neuromuscular disease is often limited due to pain, activity intolerance, musculoskeletal impairments, fatigue and other such related variables. Often, submaximal exercise testing can overcome some of these obstacles, and as such, is used frequently in the clinical environment. Non-ambulatory exercise testing utilizing an arm ergometer specifically has not been studied as heavily, especially in those with progressive myopathies. For this study, we will use maximal aerobic capacity testing for individuals with Cystinosis Myopathy utilizing a bike ergometer to allow testing of individuals regardless of their ambulatory status.

DETAILED DESCRIPTION:
High Intensity Interval Training (HIIT) has been frequently used and studied in normal populations. HIIT exercise shows improved exercise capacity with possible benefits to the neuroendocrine system and neurotransmitters associated with well-being. In this study, we plan to compare aerobic capacity changes during seated HIIT aerobic exercise of individuals with Cystinosis Myopathy. Additionally, we will assess peripheral fatigue using quantitative strength force production and slope decline before and after HIIT aerobic training.

High Intensity interval training: HIIT is a type of interval training that alternates between intense efforts and less intense recovery periods. Benefits include improved aerobic capacity, anaerobic energy, oxygen transport, lactate clearance and neuromuscular coordination. In this study, participants will train at maximal intensities (90-95% of VO2 Max) to place less strain on the neuromuscular system. The goal is to work at longer time periods above the lactate threshold causing an increase in blood lactate concentrations and improve muscles ability to oxidize fats and carbohydrates . Other studies have shown cardiovascular benefits of improved heart volume, maximal mitochondrial capacity and cardiac efficiency. HIIT training compared to regular moderate intensity exercise shows no difference in safety risk for individuals who are sedentary, have heart disease or stroke. However, compared to continuous exercise, HIIT appears to have improved oxygen consumption, blood vessel function, and glucose metabolism in healthy individuals .

Methods:

Ten participants who consent to participate in this exercise study, with no history or evidence of cardiomyopathy or conduction abnormality, and pass screening assessment for ability to complete the training program will be included and provided with an activity monitor, lower/upper extremity ergometer and remote fitness application that the participant will follow for the in-home training.

This study will be a HIIT based home exercise program where participants will perform the lower extremity ergometer based on a HIIT protocol 3x week for 20-30 minutes for a total of 8 weeks.

Baseline and end of training assessments will include MRI, muscle biopsy, strength and functional assessments including VO2 Max exercise testing and Timed Up and Go (TUG) tests. Participants will be provided hands on training to use the exercise ergometer, activity monitor, heart rate monitor, and exercise plan. The activity monitor will be programmed so that the researchers have access to monitor the patient's activity to ensure adherence to the program and changes in activity level. Additionally, a HIIT based fitness application will be installed on the participant's phone. The fitness application will be used as a guided exercise program and also allow the researchers a secondary method to monitor exercise adherence. The researchers will have access to the participant's Fitbit and fitness application use to monitor compliance. Participants who miss one session will be contacted by researchers as a reminder to follow the exercise plan. Skype sessions will be used as needed based on participant adherence or as needed for safety.

ELIGIBILITY:
Inclusion Criteria:

>=18 years -<= 60 years male or female with documented diagnosis of Cystinosis

Exclusion Criteria:

All Cystinosis participants:

* female subject who is known or suspected to be pregnant
* excluded for other illnesses or medications that may impact growth, nutritional status, development, or bone health unrelated to cystinosis

Exercise intervention:

* exercise limitation due to pre-existing heart disease
* individuals on medications that limit heart rate (beta adrenergic blockers)
* unable to plantar flex or dorsiflex ankle against resistance
* unable to use pedal ergometer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
VO2 max testing | 30-45 minutes
  Patients will undergo exercise stress testing using a recumbent cycle ergometry pre and post exercise intervention: Baseline and after week 12. We will use a ramping protocol to maintain a pedal cadence between 50-80RPM which will yield progressive workload increments of 5-10 Watts. Participants will be continuously monitored for any discomfort or pain that they may experience. Maximal effort will be verified as volitional fatigue (OMNI Scale≥8, the inability to maintain pedal cadence at 50 rpm for 10 or more seconds, and/or respiratory exchange ratio (RER; carbon dioxide production/oxygen uptake)>1.0). Standard ACSM exercise termination criteria will be applied. Measurements will end immediately following exercise. Using this method, peak oxygen uptake (VO2peak) will be identified as the highest oxygen uptake measured during exercise.

SECONDARY OUTCOMES:
Biodex Quantitative muscle testing | 30 minutes
  Biodex isokinetic dynamometer is used for testing strength throughout an entire arc of range of motion. It is commonly used to assess strength and well validated in the orthopedic field. Patients will undergo testing of both knee extensors and flexors strength as part of this protocol. Each participant will be tested in a seated position with hip flexion at 110-125 degrees; stabilization straps will be applied at the trunk and thighs. The resistance pad will be placed proximally at the medial malleolus. Range of motion at the knee will be set from 0-90 degrees. Vocal encouragement will be provided during the test and standardized for consistency between measures. Average power and H/Q ratios will be calculated and reported by the Biodex.
Timed up and Go (TUG) Test | 5 minutes
  This is a functional timed test requiring the participant to get up from a chair walk 3 meters and sit back down in the chair. It has been used to asses function and balance.
Activity Monitor | 24 hours
  We will use an activity monitor to be worn by the participant throughout the trial. For this study, participants will be issued fitbit that will estimate characteristics of physical activity. The activity monitor will help determine adherence to the exercise intervention via monitoring of the clinical research team for increased exercise at times and frequencies indicated by the protocol. Additionally, this will give us a measurable tool to assess possible changes in activity while on the study. We will compare baseline measures to changes at the end of the 12 week intervention program.
Activity Questionnaire | 5 minutes
  We will conduct a the International Physical Activity Questionnaire (IPAQ). It is developed to assess physical activity and sedentary lifestyle among people 15-69 years old. There are 5 activity domains that should be answered based on activity in the last 7 days. It has 3 categorical levels of scoring with 1 being low and 3 high. It will be provided to all participants before the start of the intervention, 8 weeks and 12 weeks. This questionnaire will help determine any changes in behavior or activity during the exercise intervention period. The questionnaire asks about amount of time the participant participates in organized sports, gym, outdoor activities, and physical exercise. This activity monitor has been used in a Cystinosis natural history study.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsampalieros A, Gupta P, Denburg MR, Shults J, Zemel BS, Mostoufi-Moab S, Wetzsteon RJ, Herskovitz RM, Whitehead KM, Leonard MB. Glucocorticoid effects on changes in bone mineral density and cortical structure in childhood nephrotic syndrome. J Bone Miner Res. 2013 Mar;28(3):480-8. doi: 10.1002/jbmr.1785. PMID 23044926
- [Background] Hafstad AD, Boardman NT, Lund J, Hagve M, Khalid AM, Wisloff U, Larsen TS, Aasum E. High intensity interval training alters substrate utilization and reduces oxygen consumption in the heart. J Appl Physiol (1985). 2011 Nov;111(5):1235-41. doi: 10.1152/japplphysiol.00594.2011. Epub 2011 Aug 11. PMID 21836050
- [Background] Hood MS, Little JP, Tarnopolsky MA, Myslik F, Gibala MJ. Low-volume interval training improves muscle oxidative capacity in sedentary adults. Med Sci Sports Exerc. 2011 Oct;43(10):1849-56. doi: 10.1249/MSS.0b013e3182199834. PMID 21448086
- [Background] Milanovic Z, Sporis G, Weston M. Effectiveness of High-Intensity Interval Training (HIT) and Continuous Endurance Training for VO2max Improvements: A Systematic Review and Meta-Analysis of Controlled Trials. Sports Med. 2015 Oct;45(10):1469-81. doi: 10.1007/s40279-015-0365-0. PMID 26243014
- [Background] Jelleyman C, Yates T, O'Donovan G, Gray LJ, King JA, Khunti K, Davies MJ. The effects of high-intensity interval training on glucose regulation and insulin resistance: a meta-analysis. Obes Rev. 2015 Nov;16(11):942-61. doi: 10.1111/obr.12317. PMID 26481101
- [Background] Helou K, El Helou N, Mahfouz M, Mahfouz Y, Salameh P, Harmouche-Karaki M. Validity and reliability of an adapted arabic version of the long international physical activity questionnaire. BMC Public Health. 2017 Jul 24;18(1):49. doi: 10.1186/s12889-017-4599-7. PMID 28738790
- [Background] Silsbury Z, Goldsmith R, Rushton A. Systematic review of the measurement properties of self-report physical activity questionnaires in healthy adult populations. BMJ Open. 2015 Sep 15;5(9):e008430. doi: 10.1136/bmjopen-2015-008430. PMID 26373402
- [Result] Wetzsteon RJ, Kalkwarf HJ, Shults J, Zemel BS, Foster BJ, Griffin L, Strife CF, Foerster DL, Jean-Pierre DK, Leonard MB. Volumetric bone mineral density and bone structure in childhood chronic kidney disease. J Bone Miner Res. 2011 Sep;26(9):2235-44. doi: 10.1002/jbmr.427. PMID 21590737